CLINICAL TRIAL: NCT02905513
Title: A Randomised Controlled Trial of an Intervention Delivered by App Instant Messaging to Increase the Acceptability of Effective Contraception Among Young People in Tajikistan
Brief Title: An Intervention Delivered by App Instant Messaging to Increase the Acceptability of Effective Contraception Among Young People in Tajikistan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: International Planned Parenthood Federation (Other); Tajik Family Planning Alliance (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 10998
Record Dates: First submitted 2016-09-14; First posted 2016-09-19 (Estimated); Last update posted 2018-02-07 (Actual); Status verified 2017-09

CONDITIONS: Contraception
Keywords: Reproductive health

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): App plus the contraceptive instant messages
  Interventions: Behavioral: Contraceptive app instant messages; Other: Mobile phone app
- Control (Placebo Comparator): App only
  Interventions: Other: Mobile phone app

INTERVENTIONS:
Behavioral: Contraceptive app instant messages
  Arms: Intervention
Other: Mobile phone app

SUMMARY:
This randomised controlled trial will establish the effect a contraceptive intervention delivered by mobile phone app instant messaging on the acceptability of effective contraception in Tajikistan. Woman and men aged 16-24 will be randomised to have access to the Tajik Family Planning Alliance's sexual and reproductive health app (control) or the app plus 0-3 instant messages a day for 4 months (intervention). Participants will complete a questionnaire at baseline and 4 months.

ELIGIBILITY:
Inclusion Criteria:

* Aged 16-24
* Own a personal Android mobile phone
* Live in Tajikistan

Exclusion Criteria:

* Cannot read Tajik or Russian

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 580 (Actual)
Dates: Start 2016-11-16 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Acceptability of at least one method of effective contraception | 4 months
  The proportion reporting that at least one method of effective contraception is acceptable (pill, intrauterine device, injection, implant)

SECONDARY OUTCOMES:
Use of effective contraception | 4 months
  The proportion reporting current use of effective contraception (pill, intrauterine device, injection, implant)
Acceptability of individual effective contraceptive methods | 4 months
  The proportion reporting that individual methods of effective contraception are acceptable (pill, intrauterine device, injection, implant)
Discontinuation of effective contraception | 4 months
  The proportion reporting use (or partner's use) of effective contraception at any time during the 4 months (pill, intrauterine device, injection, implant, patch)
Service uptake | 4 months
  The proportion reporting attending a sexual health service during the 4 months
Unintended pregnancy | 4 months
  The proportion reporting that they became pregnant (or partner became pregnant) and did not want to become pregnant during the study
Induced abortion | 4 months
  The proportion reporting having (or partner having) an abortion during the study

OTHER OUTCOMES:
Knowledge of effective contraception | 4 months
  Score on the knowledge measure
Perceived norms in relation to using and communicating with partners about contraception | 4 months
  Responses to the perceived norms scales
Personal agency in using (women only) and communicating with partners about contraception | 4 months
  Responses to the personal agency scales
Intention to use effective contraception (women only) | 4 months
  Score on the intention measure
Intervention 'dose' received | 4 months
  If participants read all, some, most or none of the messages and if they stopped the messages

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Free, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- Tajik Family Planning Alliance, Dushanbe, Tajikistan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Palmer MJ, Henschke N, Villanueva G, Maayan N, Bergman H, Glenton C, Lewin S, Fonhus MS, Tamrat T, Mehl GL, Free C. Targeted client communication via mobile devices for improving sexual and reproductive health. Cochrane Database Syst Rev. 2020 Jul 14;8(8):CD013680. doi: 10.1002/14651858.CD013680. PMID 32779730
- [Derived] McCarthy O, Ahamed I, Kulaeva F, Tokhirov R, Saibov S, Vandewiele M, Standaert S, Leurent B, Edwards P, Palmer M, Free C. A randomized controlled trial of an intervention delivered by mobile phone app instant messaging to increase the acceptability of effective contraception among young people in Tajikistan. Reprod Health. 2018 Feb 13;15(1):28. doi: 10.1186/s12978-018-0473-z. PMID 29433506
- [Derived] McCarthy O, Leurent B, Edwards P, Tokhirov R, Free C. A randomised controlled trial of an intervention delivered by app instant messaging to increase the acceptability of effective contraception among young people in Tajikistan: study protocol. BMJ Open. 2017 Sep 21;7(9):e017606. doi: 10.1136/bmjopen-2017-017606. PMID 28939582